CLINICAL TRIAL: NCT07179120
Title: Male Fertility Preservation: Efficacy Evaluation of GLP-1Receptor Agonist Therapy for Infertility in Obese Males - A Multicenter Clinical Randomized Controlled Trial
Brief Title: Can Fat-Burning Shots Boost Fertility? Comparing Weight-Loss Injections vs. Healthy Habits for Obese Men With Low Sperm Health
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-354
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Obesity-related Male Infertility
Keywords: Obesity; Male Infertility; GLP-1 Receptor Agonists; Semaglutide; Tirzepatide; Fertility Preservation; Semen Quality; Randomized Controlled Trial; Multicenter Study
MeSH Terms: conditions — Obesity; Infertility, Male | interventions — semaglutide; Tirzepatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Semaglutide Injection Therapy (Intervention A Group) (Experimental): Participants receive subcutaneous semaglutide injections titrated from 0.25mg to 1.0mg weekly over 8 weeks, maintained through week 32. Combined with standardized lifestyle intervention (identical to Control Group). Dose adjustments follow predefined tolerability criteria.
  Interventions: Drug: Semaglutide (Rybelsus®)
- Tirzepatide Injection Therapy (Intervention B Group) (Experimental): Participants receive subcutaneous tirzepatide injections titrated from 2.5mg to 15mg weekly over 12 weeks, maintained through week 32. Combined with standardized lifestyle intervention (identical to Control Group). Dose adjustments follow predefined tolerability criteria
  Interventions: Drug: Tirzepatide
- Lifestyle Modification Management (Control Group) (Experimental): Participants receive standardized intensive lifestyle intervention including personalized dietary guidance (calorie-restricted Mediterranean diet), structured aerobic/resistance exercise protocol (150 mins/week), and behavioral coaching. No pharmacotherapy is administered. Interventions are delivered through weekly sessions for first 12 weeks followed by biweekly sessions.
  Interventions: Behavioral: Standardized Lifestyle Intervention

INTERVENTIONS:
Drug: Semaglutide (Rybelsus®) — Participants receive once-weekly subcutaneous injections of Semaglutide. The dose is titrated every 4 weeks: 0.25 mg (Weeks 1-4), 0.5 mg (Weeks 5-8), and maintained at 1.0 mg from Week 9 to Week 32. Injections are administered in the abdomen, thigh, or upper arm
  Arms: Semaglutide Injection Therapy (Intervention A Group)
Drug: Tirzepatide — Participants receive once-weekly subcutaneous injections of Tirzepatide. The dose is titrated every 4 weeks: 2.5 mg (Weeks 1-4), 5 mg (Weeks 5-8), 10 mg (Weeks 9-12), and maintained at 15 mg from Week 13 to Week 32. Injections are administered in the abdomen, thigh, or upper arm
  Arms: Tirzepatide Injection Therapy (Intervention B Group)
Behavioral: Standardized Lifestyle Intervention — Participants receive individualized intensive lifestyle management, including a calorie-restricted Mediterranean diet (daily deficit of 500 kcal), structured aerobic and resistance exercise (150 mins/week), and behavioral coaching. Delivered through weekly face-to-face sessions for the first 12 weeks, followed by bi-weekly sessions for the remaining 20 weeks. No pharmacotherapy is administered.
  Arms: Lifestyle Modification Management (Control Group)

SUMMARY:
Why is this study being done? Obesity can harm men's fertility by lowering sperm quality and hormone levels, making it harder to have children. Weight loss through diet and exercise helps, but it's often hard to stick with. New medicines called GLP-1 receptor agonists, like semaglutide (Ozempic) and tirzepatide (Mounjaro), help people lose weight and improve health. Early studies suggest these drugs might also boost sperm health in obese men, but more proof is needed. This study tests if these drugs can safely improve fertility in obese men who are having trouble conceiving.

What will happen in this study?

This is a 48-week study at several hospitals in China. About 180 men will be randomly assigned to one of three groups:

Group 1: Standard lifestyle changes, like a healthy diet and exercise, guided by experts.

Group 2: Weekly injections of semaglutide, starting low and increasing as tolerated.

Group 3: Weekly injections of tirzepatide, starting low and increasing as tolerated.

All men will have regular check-ups, including blood tests, semen analysis, and weight measurements. We will track sperm quality, hormone levels, weight loss, and whether their partners get pregnant naturally. The study includes an 8-week adjustment period, 24 weeks of treatment, and 16 weeks of follow-up.

Who can join this study? Men aged 20-45 who are married, obese (BMI 28 or higher or waist size 90 cm or more), and have been trying to have a baby for at least a year without success due to low sperm count or poor sperm movement. Their female partners must be under 40 and have no major fertility issues. Men must be willing to attend visits and provide samples. People with serious health problems, recent use of similar drugs, or other causes of infertility (like genetic issues) cannot join.

How long will this study last? The full study lasts 48 weeks (about 11 months), with visits every 4-8 weeks, plus monthly phone check-ins for pregnancy updates.

What are the possible benefits and risks? Benefits: If the drugs work, men may lose weight, improve sperm quality, and have a better chance of their partners getting pregnant naturally. They might also feel healthier overall. Risks: Common side effects include nausea, vomiting, or diarrhea from the drugs, which usually improve over time. Rare risks include pancreas inflammation or gallbladder issues. Lifestyle changes might cause minor injuries from exercise. All side effects will be monitored closely, and participants can quit anytime. Insurance covers any study-related harm.

ELIGIBILITY:
Inclusion Criteria:

* (1) Married men aged 20-45 (considering childbearing age and ensuring fertility requirements), with female spouses <40 years old and no significant infertility factors.

  (2) Meeting China's adult obesity criteria: BMI ≥28 kg/m² or meeting central obesity criteria (waist circumference ≥90 cm).

  (3) Meeting WHO diagnostic criteria for male infertility: Failure to achieve pregnancy after ≥1 year of unprotected normal sexual activity, diagnosed as male-factor infertility after basic evaluation (e.g., oligospermia, asthenospermia, or high sperm deformity rate; excluding azoospermia), with essentially normal fertility function in the female spouse.

  (4) Abnormal semen analysis: Baseline semen testing shows low sperm concentration or motility (e.g., sperm concentration <15×10⁶/mL or progressive motility <32%).

  (5) Willing to undergo randomization and corresponding interventions, able to attend regular follow-ups, and provide semen and blood samples.

  (6) Informed consent to participate in the study and signing of the informed consent form.

Exclusion Criteria:

* (1) Other clear causes affecting male fertility: e.g., obstructive azoospermia, severe oligospermia (sperm concentration <5×10⁶/mL), history of bilateral cryptorchidism surgery, genetic abnormalities (chromosomal anomalies such as Klinefelter syndrome, Y-chromosome microdeletions), severe reproductive tract damage, or infection history.

  (2) Spouse has significant infertility factors (e.g., bilateral tubal blockage, severe ovulation disorders) without effective treatment, which may severely impact pregnancy outcomes.

  (3) Previous bariatric surgery (e.g., gastric bypass, sleeve gastrectomy) or current use of other weight-loss medications (e.g., orlistat), or weight fluctuation >5% within 3 months before enrollment.

  (4) Endocrine diseases affecting reproduction or sexual function: e.g., uncontrolled diabetes (HbA1c >9%) or insulin-treated diabetes, clinically significant thyroid dysfunction, hyperprolactinemia.

  (5) Severe systemic diseases: Including significant cardiovascular diseases (unstable angina, class III-IV heart failure, etc.), active liver disease (transaminases >2× upper limit of normal), severe renal impairment (eGFR <30 mL/min/1.73m²), etc., making participation in clinical trials inappropriate.

  (6) History of acute pancreatitis; personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2) (GLP-1RA is contraindicated in these cases)

  ; or conditions unsuitable for weight-loss medications, such as severe hepatic/renal impairment or gallstones.

  (7) Use of GLP-1 receptor agonist therapy within the past 6 months. (8) Received other fertility-improving treatments within the past 6 months that cannot be discontinued (e.g., gonadotropins, clomiphene, testosterone preparations, or other drugs affecting semen such as exogenous testosterone or 5-alpha-reductase inhibitors).

  (9) Alcohol or drug abuse. (10) Psychiatric or cognitive disorders preventing cooperation with follow-up. (11) Any other condition deemed by the investigator to interfere with trial results or increase participant risk.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-08-12 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Sperm Concentration (million/mL) at Week 32 of Intervention | Baseline and Week 32
  Sperm concentration is measured by standardized laboratory analysis of semen samples. Values are reported in million sperm cells per milliliter (million/mL). Higher values indicate better spermatogenesis function. The World Health Organization (WHO) reference lower limit for normal concentration is ≥15 million/mL. Change is calculated as: (Week 32 value - Baseline value)

SECONDARY OUTCOMES:
Change from Baseline in Total Sperm Count at Week 32 | Baseline and Week 32
  Total sperm count is calculated from semen volume and sperm concentration. Values are reported in millions. Higher values indicate better spermatogenesis function.
Change from Baseline in Sperm Motility (Progressive + Non-progressive) at Week 32 | Baseline and Week 32
  Sperm motility assesses the percentage of sperm moving (progressive + non-progressive). Values range from 0% to 100%. Higher percentages indicate better sperm function.
Change from Baseline in Serum Total Testosterone Level at Week 32 | Baseline and Week 32
  Serum total testosterone is measured via chemiluminescence immunoassay. Reported in nanomoles per liter (nmol/L). Normal adult male range is typically 10-35 nmol/L.
Change from Baseline in Follicle-Stimulating Hormone (FSH) Level at Week 32 | Baseline, Week 32
  Serum FSH concentration is measured by chemiluminescence immunoassay, reported in international units per liter (IU/L). It assesses pituitary-gonadal axis function. Normal reference range for adult males is typically 1.5-12.4 IU/L.
Change from Baseline in Luteinizing Hormone (LH) Level at Week 32 | Baseline, Week 32
  Serum LH concentration is measured by chemiluminescence immunoassay, reported in international units per liter (IU/L). It assesses pituitary-gonadal axis function. Normal reference range for adult males is typically 1.7-8.6 IU/L.
Change from Baseline in Body Mass Index (BMI) at Week 32 | Baseline, Week 16, Week 32
  Body weight is measured using a calibrated digital scale, reported in kilograms (kg). Change is calculated as post-intervention value minus baseline value. A negative value indicates weight loss.
Change from Baseline in Waist Circumference at Week 32 | Baseline, Week 16, Week 32
  Waist circumference is measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest using a non-elastic tape, reported in centimeters (cm). It assesses central obesity. A value ≥90 cm in Asian males indicates increased health risk.
Number of Participants Achieving Natural Pregnancy Within 48 Weeks | Monthly during the study, up to Week 48
  Natural pregnancy is confirmed by a positive serum β-hCG test (>5 mIU/mL) followed by transvaginal ultrasound verification of an intrauterine gestational sac. It is reported as a binary outcome (Yes/No) for each participant.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0 | From first dose until 30 days after last dose (up to Week 48+30)
  All adverse events occurring after the initiation of treatment are assessed by the investigator for severity (Grade 1-5 Mild to Death) and relationship to study intervention according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

IPD SHARING:
Plan to Share IPD: No